CLINICAL TRIAL: NCT03429205
Title: The Efficacy of External Warming During Laparoscopic Bariatric Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting pace too slow.
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, David Goitein MD, Director, Bariatric and Metabolic Surgery, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4578-17-SMC
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hypothermia; Morbid Obesity; Bariatric Surgery Candidate
Keywords: Sleeve gastrectomy; Roux-Y gastric bypass; Single anastomosis gastric bypass; Hypothermia; External heating blanket
MeSH Terms: conditions — Hypothermia; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No heating - Study group (Experimental): Patient will undergo bariatric surgery without utilization of external heating device.
  Interventions: Other: No external heating used during surgery
- Heating - Control group (Other): Patient will undergo bariatric surgery with utilization of external heating device.
  Interventions: Other: External heating blanket used during surgery

INTERVENTIONS:
Other: No external heating used during surgery — Deviation from external heating for all surgery standard
  Arms: No heating - Study group
Other: External heating blanket used during surgery — Standard external heating plan used in all surgery types
  Arms: Heating - Control group

SUMMARY:
External warming is routinely used in general surgery to offset the deleterious effects of hypothermia. It entails deployment of a disposable, external heating blanket attached to a regulated hot-air pump.

The need for external warming in the morbidly obese population undergoing short laparoscopic procedures is unclear. If proven to be unnecessary, time and momentary costs could be lowered.

The study will compare core-temperature dynamics during laparoscopic bariatric procedures anticipated to last <2h. The study group will be left without a warming blanket while the control group will receive routine external warming. Post-anesthesia care unit (PACU) arrival temperature will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for bariatric surgery
* Surgery time estimated to be < 2 hours

Exclusion Criteria:

* Previous abdominal surgeries (except laparoscopic cholecystectomies, appendectomies and hysterectomies+/-oophorectomies).
* Surgery time estimated to be more than 2 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Intraoperative core-temperature decline | Surgery duration, up to 2 hours from surgery start-time
  Core-temperature will be continuously measured throughout surgery
Arrival temperature at post anesthesia care unit (PACU) | arrival to recovery room, up to 2 h from surgery start-time
  Core temperature upon arrival to recovery room

SECONDARY OUTCOMES:
Hypothermia events | 3 hours from surgery start-time
  Measurement of core temperature <35 C
Intraoperative blood loss | Surgery duration, up to 2 hours from surgery start-time
  Intraoperative bleeding score will be used
Post operative complications | 30 days postoperatively
  Complications after surgery (30 days), graded according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No